CLINICAL TRIAL: NCT07022223
Title: A Single-arm, Prospective Clinical Study to Evaluate the Efficacy and Safety of Orelabrutinib Combined With Rituximab as First-line Systemic Treatment for Marginal Zone Lymphoma
Brief Title: Orelabrutinib Combined With Rituximab as First-line Systemic Treatment for Marginal Zone Lymphoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: The Second Affiliated Hospital of Jiaxing University (Other); Taizhou First People's Hospital (Other); Huzhou Central Hospital (Other); Zhejiang Cancer Hospital (Other); Dongyang People's Hospital (Other); Yuyao People's Hospital (Other); Taizhou Hospital (Other); Shaoxing Central Hospital (Other); Affiliated Hospital of Jiaxing University (Other); Shaoxing People's Hospital (Other); Taizhou Hospital of Zhejiang Province affiliated to Wenzhou Medical University (Other); The Central Hospital of Lishui City (Other); Second Affiliated Hospital of Wenzhou Medical University (Other); Ningbo People's Hospital (Unknown); The People's Hospital of Quzhou (Other); Zhejiang University (Other); Zhuji People's hospital (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-1336
Record Dates: First submitted 2025-06-01; First posted 2025-06-15 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-03

CONDITIONS: Marginal Zone Lymphoma(MZL)
MeSH Terms: conditions — Lymphoma, B-Cell, Marginal Zone

STUDY DESIGN:
Intervention Model Description: Orelabrutinib combined with rituximab regimen
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- orelabrutinib combined with rituximab regimen (Experimental): All participants will receive induction therapy with the orelabrutinib and rituximab regimen. The treatment cycle is 28 days, with a total of 6 cycles. The induction treatment period is as follows:
  Cycle 1: Rituximab, 375 mg/m², on Day 1. Cycles 2-6:Orelabrutinib, 150 mg, once daily orally, from Day 1 to Day 28. Rituximab, 375 mg/m², on Day 1.
  Patients who achieve a partial response (PR) or better will enter a 2-year maintenance period with orelabrutinib.
  Interventions: Drug: orelabrutinib combined with rituximab regimen

INTERVENTIONS:
Drug: orelabrutinib combined with rituximab regimen — All participants will receive induction therapy with the orelabrutinib and rituximab regimen. The treatment cycle is 28 days, with a total of 6 cycles. The induction treatment period is as follows:
  Cycle 1: Rituximab, 375 mg/m², on Day 1. Cycles 2-6:Orelabrutinib, 150 mg, once daily orally, from Day 1 to Day 28. Rituximab, 375 mg/m², on Day 1.
  Patients who achieve a partial response (PR) or better will enter a 2-year maintenance period with orelabrutinib.

SUMMARY:
This is a single-arm, prospective clinical study to evaluate the efficacy and safety of orelabrutinib combined with rituximab as first-line systemic treatment for marginal zone lymphoma.

DETAILED DESCRIPTION:
Marginal zone lymphoma (MZL) is a relatively common type of B-cell non-Hodgkin lymphoma (B-NHL), with an incidence rate second only to diffuse large B-cell lymphoma (DLBCL) and follicular lymphoma (FL). The Bruton tyrosine kinase (BTK) signaling pathway plays a significant role in B-cell malignancies. Most B-cell malignancies require activation of the B-cell receptor (BCR), and BTK, located downstream of the BCR, plays a crucial role in B-cell proliferation, apoptosis, differentiation, and migration induced by antigens. Currently, there is no unified treatment regimen with high-level evidence for the treatment of newly diagnosed MZL. As mentioned above, although high-intensity immunochemotherapy regimens achieve high response rates and durable remission, they also bring higher treatment-related safety risks (with a rate of grade 3 or higher adverse events of about 80%), including treatment-related deaths. Therefore, exploring effective chemotherapy-free regimens for MZL patients is a scientifically valuable and clinically meaningful attempt. Drugs such as BTK inhibitors and CD20 monoclonal antibodies have shown good therapeutic activity and clinical data as single agents. This is a single-arm, prospective clinical study to evaluate the efficacy and safety of orelabrutinib combined with rituximab as first-line systemic treatment for marginal zone lymphoma. All subjects will receive induction treatment with the orelabrutinib and rituximab regimen. The treatment cycle is 28 days, with a total of 6 cycles. Patients who achieve a partial response (PR) or better will enter a 2-year maintenance period with orelabrutinib.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years, regardless of gender;
* Histologically confirmed CD20-positive marginal zone lymphoma, including MALT, SMZL, and NMZL, with at least one lesion outside the spleen measuring more than 1.5 cm in any axis;
* MZL that has progressed or relapsed after prior local therapy (including surgery, radiotherapy, anti-Helicobacter pylori treatment, and anti-hepatitis C treatment), or is not suitable for local therapy;
* ECOG performance status of 0-2;
* Presence of an indication for treatment as judged by the investigator (symptomatic, cytopenia, risk of end-organ damage, bulky disease, ongoing progression, or patient's desire for treatment);
* Adequate function of major organs, as follows:
* Hematology: Absolute neutrophil count ≥ 1.5×109/L, platelets ≥ 75×109/L, hemoglobin ≥ 75 g/L; if there is bone marrow involvement, absolute neutrophil count ≥ 1.0×109/L, platelets ≥ 50×109/L, hemoglobin ≥ 50 g/L;
* Biochemistry: Total bilirubin ≤ 1.5 times the upper limit of normal (ULN), AST or ALT ≤ 2 times ULN; serum creatinine ≤ 1.5 times ULN; serum amylase ≤ ULN;
* Coagulation: International normalized ratio (INR) ≤ 1.5 times ULN.
* Life expectancy of ≥ 3 months;
* Voluntary written informed consent obtained before screening for the trial.

Exclusion Criteria:

* Currently or previously having other malignancies, unless there is evidence of no recurrence or metastasis within the past 5 years after curative treatment;
* Lymphoma involvement of the central nervous system or transformation to high-grade lymphoma;
* Non-hematological toxicities from prior anti-cancer treatments not recovered to ≤ Grade 1 (excluding alopecia);
* Presence of uncontrolled or significant cardiovascular disease, including:
* New York Heart Association (NYHA) Class II or higher congestive heart failure, unstable angina, myocardial infarction within 6 months before the first administration of the study drug, or arrhythmias requiring treatment at screening, left ventricular ejection fraction (LVEF) < 50%;
* Primary cardiomyopathy (such as dilated cardiomyopathy, hypertrophic cardiomyopathy, arrhythmogenic right ventricular cardiomyopathy, restrictive cardiomyopathy, unclassified cardiomyopathy);
* History of clinically significant QTc interval prolongation, or QTc interval > 470 ms for females, > 450 ms for males during the screening period;
* Symptomatic or medically treated coronary artery disease;
* Uncontrolled hypertension (defined as blood pressure not reaching target levels despite a reasonable and tolerable full dose of three or more antihypertensive drugs (including diuretics) for more than one month, or requiring four or more antihypertensive drugs to effectively control blood pressure).
* Active bleeding within 2 months before screening, or currently taking anticoagulant drugs, or deemed by the investigator to have a clear tendency to bleed;
* Urine protein ≥ 2+, and 24-hour urine protein quantification ≥ 2 g/24 hours;
* History of deep vein thrombosis or pulmonary embolism within the past six months;
* History of organ transplantation or allogeneic bone marrow transplantation;
* Major surgery within 6 weeks before screening or minor surgery within 2 weeks before screening. Major surgery is defined as surgery using general anesthesia, but diagnostic endoscopy is not considered major surgery. Insertion of a vascular access device will be exempt from this exclusion criterion;
* Active infection or uncontrolled HBV (HBsAg positive and/or HBcAb positive with positive HBV DNA titer), HCV Ab positive, HIV/AIDS, or other severe infectious diseases;
* Currently having pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, radiation pneumonitis, drug-related pneumonia, or other conditions that significantly affect pulmonary function;
* Previous treatment with BTK, BCR pathway inhibitors (such as PI3K, Syk), or BCL-2 inhibitors;
* Suitable and preparing for stem cell transplantation;
* Any psychiatric or cognitive impairment that may limit their understanding, execution of the informed consent form, and compliance with the study;
* Subjects with drug abuse or alcoholism;
* Pregnant, breastfeeding women, and fertile subjects unwilling to use contraception;
* Need to continuously take drugs with moderate to severe inhibitory or strong inducing effects on cytochrome P450 CYP3A;
* Any other condition deemed by the investigator as unsuitable for participation in this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Estimated)
Dates: Start 2025-03-11 (Actual); Primary Completion 2027-09-11 (Estimated); Study Completion 2029-09-11 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) | up to 6 months
  ORR is defined as the proportion of patients with a response of CR or PR

SECONDARY OUTCOMES:
Complete Response Rate (CR) | up to 6 months
  The rate of patients who achieved complete response after treatment
Best Overall Response (BOR) | up to 6 months
  The best response achieved by the patient from the start of treatment until disease progression or the initiation of a new treatment regimen.
Duration of Response (DoR) | Up to 2 years
  Duration of response as defined as the period from the first response (at least PR) to treatment until evidence of disease progression, relapse or death of any cause. Patients alive without progression and relapse will be censored at the latest tumor assessment date or the stopping date.
2 years progression-free survival Progression free survival | From date of signing the informed consent until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 2 years
  PFS is defined as the time from registration to the first occurrence of progression or relapse as assessed by the investigator, or death from any cause. PFS for patients without disease progression, relapse, or death will be censored at the time of the last tumor assessment
2 years overall survival | From date of signing the informed consent until the date of death from any cause, whichever came first, assessed up to 2 years
  Overall survival is defined as the period from the induction registration to death from any cause. Patients who have not died until the time of the analysis will be censored at their last contact date.
time to complete response within 24 months (TTCR24) | up to 2 years
  TTCR24 is deﬁned as the time from randomization to ﬁrst CR, and censored at 24 months
complete response (CR) at 24 months | up to 2 years
  CR24 is deﬁned as the CR rate at 24 months

CONTACTS AND LOCATIONS:
Locations (18):
- China (18):
  - Second Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang
  - Dongyang People's Hospital, Dongyang
  - Affiliated Hangzhou First People's Hospital, Hangzhou
  - Zhejiang cancer Hospital, Hangzhou
  - Huzhou Central Hospital, Huzhou
  - Affiliated Hospital of Jiaxing University, Jiaxing
  - The Second Affiliated Hospital of Jiaxing University, Jiaxing
  - Lishui central Hospital, Lishui
  - the Affiliated Peopele'S Hospital of Ningbo University, Ningbo
  - Quzhou People's Hospital, Quzhou
  - Shaoxing Central Hospital, Shaoxing
  - shaoxing People's Hospital, Shaoxing
  - Taizhou Central Hospital, Taizhou
  - Taizhou First People's Hospital, Taizhou
  - Taizhou Hospital ofzhejiang Province, Taizhou
  - The Second Affiliated Hospital and Yuying childrens Hospital of Wenzhou Medical University, Wenzhou
  - Yuyao People's Hospital, Yuyao
  - Affiliated Zhuji Hospital ofWenzhou Medical University, Zhuji